CLINICAL TRIAL: NCT04055792
Title: Sintilimab Combined With Anlotinib as Second- or Further-line Therapy for Extensive Disease Small Cell Lung Cancer: A Prospective, Single-arm, Phase II Study
Brief Title: Sintilimab Combined With Anlotinib as Second or Further-line Therapy for ED-SCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiming Wang, chief physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200526
Record Dates: First submitted 2019-08-11; First posted 2019-08-14 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Extensive Disease Small Cell Lung Cancer
Keywords: extensive disease small cell lung cancer; PD-1 inhibitor; anti-angiogenesis; second or further-line setting
MeSH Terms: conditions — Neoplasm Metastasis | interventions — sintilimab; anlotinib

STUDY DESIGN:
Intervention Model Description: A prospective, single-arm, Phase II study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab combine with Anlotinib (Experimental): Sintilimab 200 mg on day 1 and oral daily Anlotinib 12 mg on days 1-14 once every 3 weeks
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg intravenously on day 1 and Anlotinib 12 mg on days 1-14 once every 3 weeks
  Other Names: Anlotinib

SUMMARY:
Small cell lung cancer (SCLC) accounts for 10-15% of lung cancer. More than 70% of SCLC patients are diagnosed with advanced stage (ED-SCLC) at diagnosis. ED-SCLC is highly chemo-sensitive, the first-line treatment is platinum-containing double-drug chemotherapy. Although ED-SCLC is highly sensitive to chemotherapy and the objective response rate (ORR) of first-line chemotherapy is as high as 60-80%, the progression-free survival (PFS) is very short, and there is a lack of effective second-line treatment. The median overall survival (OS) of patients is only 10 months, and the 2-year survival rate is about 6%.

DETAILED DESCRIPTION:
In August 2018, the FDA approved Nivolumab as a third-line treatment for ED-SCLC patients. Sintilimab is another PD-1 inhibitor produced by China and has been approved by cFDA for lymphoma. Anlotinib is a novel multi-target tyrosine kinase inhibitor (TKI) with effect of anti-tumor angiogenesis and tumor growth inhibition. The results of ALTER1202 showed that compared with placebo, Anlotinib single-agent as third-line treatment in ED-SCLC was effective, the median PFS was 4.1 versus 0.7 months, respectively (P < 0.001).

Immunotherapy combined with anti-angiogenic therapy has been proven effective and tolerable in non-small cell lung caner (NSCLC), while its efficacy and safety in SCLC has not been reported. Therefore, the investigators conduct this study to evaluate the efficacy and safety of Sintilimab combined with Anlotinib as second or further-line therapy for ED-SCLC patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be enrolled:

* Histologically or cytologically confirmed ED-SCLC according to the VALG staging system, and not suitable for local treatment.
* Progressed after at least one line of platinum-containing chemotherapy.
* ≥1 measurable lesions based on Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST v1.1).
* Previous radiotherapy was allowed, but the radiotherapy area must be <25% of the bone marrow area (Cristy and Eckerman 1987) and no total pelvic or chest irradiation was used; the previous radiotherapy must have been completed for at least 4 weeks before the start of study drugs treatment, and the acute toxicity must have been restored; radiotherapy of local lesions cannot be included in measurable lesions unless significant progression is noted after radiotherapy.
* Prior surgery was allowed, provided that the treatment was completed at least 4 weeks before the start of study drugs treatment, and the acute toxicity must have been restored.
* ≥18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
* Life expectancy > 12 weeks.
* Adequate bone marrow, hepatic and renal function.
* Systolic blood pressure ≤160mmHg and diastolic pressure ≤90mmHg within 7 days before enrollment.
* Patients must sign study specific informed consent before registration.
* Female patients should be surgically sterilized, postmenopausal, or consent to use a medically approved contraceptive method (such as an IUD, contraceptive pill, or condom) during the study treatment period and for 6 months after the end of the study treatment period; Serum or urine pregnancy tests must be negative within 7 days prior to study enrollment and must be non-lactating; Male patients should be surgically sterilized or who have consented to use a medically approved form of contraception during the study treatment period and for 6 months after the end of the study treatment period.

Exclusion Criteria:

Any of the following conditions should not be included in this study:

* Patients with brain metastasis. Patients suspected of having brain metastases should be examined by brain CT or MRI before enrollment; Patients with a history of brain metastases must have completed treatment and no longer need corticosteroids; For asymptomatic patients, the investigator will determine whether to enroll.
* Patients with meningeal metastasis.
* Prior treatment with PD-1 inhibitor, PD-L1 inhibitor, CTLA4 inhibitor, or anti-angiogenic treatment.
* Accept any other anti-tumor treatment simultaneously.
* Diagnosed with active autoimmune diseases (congenital or acquired, patients with completely relieved or childhood vitiligo can be enrolled; patients with hypothyroidism and only need hormone replacement therapy can be rerolled; Patients with type 1 diabetes can also be enrolled).
* Diagnosed with interstitial pneumonia.
* Patients with hemorrhage tendency including acute hemorrhage of digestive tract, continuous hemorrhage disease or coagulation function disorder disease.
* Patients are using warfarin, heparin or aspirin (>325 mg/day) or NSAIDS to inhibit platelet function within 10 days prior to enrollment, or receiving dipyridamole, ticlopidine, clopidogrel or cilostazol treatment.
* Patients with accompanying diseases that seriously endanger the safety of the patient or affect the patient's completion of the study.
* Pregnant or lactating female.
* Prior other malignant diseases, except for cervical carcinoma in situ, papillary thyroid carcinoma, or non-melanoma skin cancer.
* Allergy to any component of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
PFS | 8 months
  progression free survival

SECONDARY OUTCOMES:
OS | 24 months
  overall survival
ORR | 8 months
  objective response rate
DCR | 8 months
  disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Qiming Wang, Principal Investigator — 127 Dongming Road, Zhengzhou, 450008, People's Republic of China
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma S, He Z, Liu Y, Wang L, Yang S, Wu Y, Chen H, Wu Y, Wang Q. Sintilimab plus anlotinib as second or further-line therapy for extensive disease small cell lung cancer: a phase 2 investigator-initiated non-randomized controlled trial. EClinicalMedicine. 2024 Mar 14;70:102543. doi: 10.1016/j.eclinm.2024.102543. eCollection 2024 Apr. PMID 38516099